Official Title of the study:

Fibrinolysis Compared to Thoracoscopy for Pleural Infection

NCT number:

NCT03468933

Date of the document:

July 1, 2017

## Statistical Analysis

We believe that a difference of 2 days in the length of the postintervention hospital stay between the two treatment arms would be clinically important. This rationale is based on a previous randomized study that compared VATS and streptokinase therapy in empyema (1). In that study, the number of chest tube days after VATS was  $5.8\pm1.1$  days, as compared with  $9.8\pm1.3$  days in the streptokinase group. Furthermore, a case series from MT trials reported an average postoperative stay of 7–8 days (2-5), as compared with an average of 10–13 days in IPFT trials (6,7). According to a two-sided type I error of 0.05 and 80% power, the sample size was 16 patients in each group.

All analyses were performed using GraphPad Prism (version 7.0; GraphPad Software). Descriptive statistics were used to summarize the patients' characteristics. The t test was used to examine differences between groups with parametric data and the Mann-Whitney U test was used for nonparametric data. Fisher's exact test was used for categorical variables. A P value of <0.05 was considered statistically significant.

- 1-Majid A, Kheir F, Folch A, Fernandez-Bussy S, Chatterji S, Maskey A, et al. Concurrent intrapleural instillation of tissue plasminogen activator and DNase for pleural infection: a single-center experience. Ann Am Thorac Soc 2016;13:1512–1518.
- 2-BrutscheMH, Tassi GF,Gyo" rik S,Go" keimenM, Renard C,MarchettiGP, et al. Treatment of sonographically stratified multiloculated thoracic empyema by medical thoracoscopy. Chest 2005;128:3303–3309.
- 3-Ravaglia C, Gurioli C, Tomassetti S, Casoni GL, Romagnoli M, Gurioli C, et al. Is medical thoracoscopy efficient in the management of multiloculated and organized thoracic empyema? Respiration 2012; 84:219–224.
- 4-Sole`r M, Wyser C, Bolliger CT, Perruchoud AP. Treatment of early parapneumonic empyema by "medical" thoracoscopy. Schweiz Med Wochenschr 1997;127:1748–1753.
- 5-Hardavella G, Papakonstantinou NA, Karampinis I, Papavasileiou G, Ajab S, Shafaat M, et al. Hippocrates quoted "if an empyema does not rupture, death will occur": is medical thoracoscopy able to make it rupture safely? J Bronchology Interv Pulmonol 2017;24: 15–20.
- 6-Maskell NA, Davies CW, Nunn AJ, Hedley EL, Gleeson FV, Miller R, et al.; First Multicenter Intrapleural Sepsis Trial (MIST1) Group. U.K. Controlled trial of intrapleural streptokinase for pleural infection. N Engl J Med 2005;352:865–874.

7- Rahman NM, Maskell NA, West A, Teoh R, Arnold A, Mackinlay C, et al. Intrapleural use of tissue plasminogen activator and DNase in pleural infection. N Engl J Med 2011;365:518–526.